CLINICAL TRIAL: NCT04918537
Title: Analysis of Microbiota Variations in Industry Workers Working Different Shifts and Impact of a Nutritional Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sophie Bucher Della Torre (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Sophie Bucher Della Torre, Professor Assistant, School of Health Sciences Geneva
Organization: School of Health Sciences Geneva (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: G700136106018
Record Dates: First submitted 2021-06-02; First posted 2021-06-09 (Actual); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Dysbiosis
Keywords: Gut microbiota
MeSH Terms: conditions — Dysbiosis

STUDY DESIGN:
Intervention Model Description: 3 weeks of observation 3 weeks of intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention walnuts (Experimental): During the 3 last weeks of the study, the participants will eat a 30g daily walnut serving
  Interventions: Dietary Supplement: Walnuts

INTERVENTIONS:
Dietary Supplement: Walnuts — 30g of plain walnuts in addition to habitual food intakes

SUMMARY:
Shift workers are a growing population. It is well established that these workers face an increased risk of developing chronic diseases, but the underlying mechanisms remain debated. Various factors such as internal circadian desynchronization, unhealthy lifestyle behaviours, and lack of sleep interact in complex ways. Recently, it has been suggested that the gut microbiota (GM) may play an important role in this increased risk.

The goal of this study is to describe the variations of the GM composition in shift workers across three different rotating weekly shifts (morning, afternoon, night) and to measure the impact of a 3- week walnuts supplementation intervention consisting in a controlled experimental study.

Therefore, we propose a 6-weeks study including an observational and an experimental part. First, in the observational part, we will compare the gut microbiota of shift workers across three shifts (morning, afternoon and night). In the second part of the study, participants will add to their usual intakes a daily serving of nuts (30g). Again, we will compare the gut microbiota composition across the three types of shifts. During the study, participants will record their food intake, sleep and defecation time. We will also monitor their blood glucose levels continuously during the 4 first weeks of the study.

ELIGIBILITY:
Inclusion Criteria:

* Working 3x8 shifts (weekly rotations between AM, PM and N shifts) for at least 3 months prior to the study
* No anticipated changes in shift work planning
* No prebiotics or probiotics supplements.

Exclusion Criteria:

* Antibiotic and/or immunomodulator use in the last 3 months or during the study
* Change in medication during the last month or during study
* Inflammatory bowel disease or important gut surgery
* Nuts allergy
* Major digestive tract surgery.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota composition between the first and last day of each type of shift (observation phase) | 3 weeks (6 measurements over time)
  Change in relative abundance of bacteria phyla between the first and last day of each type of shift (AM, PM, N). Assessed by 16S rRNA sequencing approach.
Change in gut microbiota composition between the first and last day of each type of shift (observation vs intervention) | 6 weeks (12 measurements over time)
  Change in relative abundance of bacteria phyla between the first and last day of each type of shift (AM, PM, N). Assessed by 16S rRNA sequencing approach.

SECONDARY OUTCOMES:
Area under the blood glucose curve between each type of shift | 3 weeks
  Area under the blood glucose curve between each type of shift (AM, PM, N). Measured using a continuous glucose monitoring.
Area under the blood glucose curve in AM shift (observation vs intervention) | week 1 vs 4
  Area under the blood glucose curve during the morning shift (AM) during the observation and the intervention. Measured using a continuous glucose monitoring.

OTHER OUTCOMES:
Mean weekly frequency of defecation between each type of shift | 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Sciences Geneva, Geneva, Carouge, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measure will be made available.
Time Frame: Data will be available within 12 months of study completion
Access Criteria: At the end of the project the data will be deposited in the Yareta repository developed by the University of Geneva OR in an institutional repository. This choice will ensure that data is archived and shared in accordance with FAIR principles.